CLINICAL TRIAL: NCT04600063
Title: Randomized Controlled Phase II Study of Isolation Procedure Versus Conventional Procedure in Distal Pancreatosplenectomy for Pancreatic Cancer
Brief Title: Isolation Procedure vs. Conventional Procedure During Distal Pancreatectosplenectomy for Pancreatic Cancer
Acronym: ISOP-DP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Director, Principal Investigator, Professor of Second Department of Surgery, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2986
Record Dates: First submitted 2020-10-18; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Resectable Pancreatic Body/Tail Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional procedure (Other): In the conventional procedure group, first, the pancreatic body and tail and spleen are mobilized (mandatory procedure), and the regional lymph nodes of the body and tail of the pancreas, such as the hepatoduodenal mesentery (No12 lymph node) and the common hepatic artery perimeter (No8), are removed. (Recommended procedure) and dissection of lymph nodes (No14p) around SMA (Recommended procedure), and after dissection of the gastro-splenic ligament and pancreas, transection of the splenic vein at the end of the resection procedure (required procedure) . However, in order to prevent bleeding and secure a safe field of view, early pancreatotomy is allowed.
  Interventions: Procedure: Isolation procedure (RAMPS procedure); Procedure: Conventional procedure
- Isolation procedure (RAMPS procedure) (Experimental): In the Isolation procedure group, the transection of the root of the splenic artery and the pancreatic transection are performed first, followed by the transection of the splenic vein (mandatory procedure). At that time, the branch from the splenic artery (dorsal pancreatic artery), the branch to the splenic vein (left gastric vein, inferior mesenteric vein), and short gastric arteriovenous are also disconnected as soon as possible (recommended procedure). An operation to lift up the pancreatic neck from the dorsal portal vein or superior mesenteric artery to expose the splenic vein (so-called tunneling) is allowed. After that, lymph node dissection such as hepatoduodenal mesentery (No12), common hepatic artery perimeter (No8), lymph node dissection around SMA (No14p) was performed (recommended procedure), and at the end of the resection operation, the pancreas body/tail and spleen are mobilized and removed (required procedure).
  Interventions: Procedure: Isolation procedure (RAMPS procedure); Procedure: Conventional procedure

INTERVENTIONS:
Procedure: Isolation procedure (RAMPS procedure) — In the Isolation procedure group, the transection of the root of the splenic artery and the pancreatic transection are performed first, followed by the transection of the splenic vein (mandatory procedure). At that time, the branch from the splenic artery (dorsal pancreatic artery), the branch to the splenic vein (left gastric vein, inferior mesenteric vein), and short gastric arteriovenous are also disconnected as soon as possible (recommended procedure). An operation to lift up the pancreatic neck from the dorsal portal vein or superior mesenteric artery to expose the splenic vein (so-called tunneling) is allowed. After that, lymph node dissection such as hepatoduodenal mesentery (No12), common hepatic artery perimeter (No8), lymph node dissection around SMA (No14p) was performed (recommended procedure), and at the end of the resection operation, the pancreas body/tail and spleen are mobilized and removed (required procedure).
Procedure: Conventional procedure — In the conventional procedure group, first, the pancreatic body and tail and spleen are mobilized (mandatory procedure), and the regional lymph nodes of the body and tail of the pancreas, such as the hepatoduodenal mesentery (No12 lymph node) and the common hepatic artery perimeter (No8), are removed. (Recommended procedure) and dissection of lymph nodes (No14p) around SMA (Recommended procedure), and after dissection of the gastro-splenic ligament and pancreas, transection of the splenic vein at the end of the resection procedure (required procedure) . However, in order to prevent bleeding and secure a safe field of view, early pancreatotomy is allowed.

SUMMARY:
In the distal pancreatectomy (including pancreatic tail resection) for invasive ductal carcinoma of the pancreas, we evaluate the usefulness of a procedure of firstly transection of splenic arteries and veins (the isolation procedure group) compared to a conventional procedure of transection of the splenic vein at the end.

ELIGIBILITY:
Inclusion Criteria:

* Resectable pancreatic cancer (Adenocarcinoma, adenosquamous cell carcinoma, mucinous carcinoma, and anaplastic carcinoma according to the 7th edition of the regulations for handling pancreatic cancer)
* ASA-PS (American Society of Anesthesiology, General condition classification) is Class 1-3.
* Age are over 20 years old.
* Able to understand the content of the research and has obtained written consent from the person himself/herself.

Exclusion Criteria:

* Non-resectable pancreatic cancer by image diagnosis at the initial diagnosis
* Cases suspected of portal vein (superior mesenteric vein) invasion
* Patients with severe ischemic heart disease
* Patients with cirrhosis or active hepatitis requiring treatment
* Patients with dyspnea requiring oxygen administration
* Patients undergoing dialysis due to chronic renal failure
* Cases in which arterial reconstruction of the superior mesenteric artery, common hepatic artery, celiac artery, etc. is considered necessary
* Patients with strong suspected paraaortic lymph node metastasis
* Active double cancer thought to affect adverse events and prognosis
* Long-term oral steroids that may affect adverse events
* Patients who are considered to have difficulty participating in the study due to psychosis or psychiatric symptoms.
* Cases other than invasive pancreatic ductal carcinoma by preoperative biopsy. Invasive intraductal papillary mucinous carcinoma (IPMC) is excluded.
* Patients who cannot use both iodine drugs and gadnium drugs due to severe drug allergy
* Cases where the prescribed procedure is difficult due to history of upper abdominal surgery such as stomach, spleen, kidney, liver, transverse colon, retroperitoneum including pancreas and pancreatitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival | Up to 24 months
  Until 2 years after last entry case undergo surgery

CONTACTS AND LOCATIONS:
Locations (10):
- Japan (10):
  - Kobe University, Kobe, Hyōgo
  - Nara Medical University, Kashihara, Nara
  - Kinki University, Sayama, Osaka
  - Osaka University, Suita, Osaka
  - Shiga Medical University, Ōtsu, Shiga
  - Kumamoto University, Kumamoto
  - Osaka City University, Osaka
  - Jikei University, Tokyo
  - Toyama University, Toyama
  - Second Department of Surgery, Wakayama Medical University, School of Medicine, 811-1 Kimiidera, Wakayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okada KI, Kawai M, Hirono S, Sho M, Tani M, Matsumoto I, Yamada S, Amano R, Toyama H, Yamashita YI, Gocho T, Shibuya K, Nagai M, Maehira H, Kamei K, Ohira G, Shirai Y, Takami H, Kimura N, Fukumoto T, Baba H, Kodera Y, Nakao A, Shimokawa T, Katsuda M, Yamaue H. ISOlation Procedure vs. conventional procedure during Distal Pancreatectomy (ISOP-DP trial): study protocol for a randomized controlled trial. Trials. 2021 Sep 16;22(1):633. doi: 10.1186/s13063-021-05523-y. PMID 34530885